CLINICAL TRIAL: NCT00689065
Title: A Phase I, Dose-Escalating Study of the Safety of Intravenous CALAA-01 in Adults With Solid Tumors Refractory to Standard-of-Care Therapies
Brief Title: Safety Study of CALAA-01 to Treat Solid Tumor Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Calando Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALAA-01-ST-001
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Cancer; Solid Tumor
Keywords: siRNA; RNA interference (RNAi); Cyclodextrin; Cancer; Neoplasms; Solid Tumor; Ovarian Cancer; Lung Cancer; Non Small Cell Lung Cancer; Pancreatic Cancer; Breast Cancer; Colon Cancer; Endometrial Cancer; Kidney (Renal Cell) Cancer; Melanoma; Prostate Cancer; Skin Cancer; Thyroid Cancer; Solid Malignancies
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Breast Neoplasms; Colonic Neoplasms; Endometrial Neoplasms; Carcinoma, Renal Cell; Melanoma; Prostatic Neoplasms; Skin Neoplasms; Thyroid Neoplasms | interventions — CALAA-01

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CALAA-01 (Experimental)
  Interventions: Drug: CALAA-01

INTERVENTIONS:
Drug: CALAA-01 — Subjects with solid tumors who satisfy the eligibility criteria will receive two, 21-day cycles of CALAA-01. A cycle will consist of four (4) 30-minute intravenous infusions administered on days 1, 3, 8, and 10 followed by 11 days of rest. If safe, a second 21-day cycle will be administered consisting of infusions on days 22, 24, 29 and 31 followed by 11 days of rest.

SUMMARY:
Rationale: CALAA-01 is a targeted therapeutic designed to inhibit tumor growth and/or reduce tumor size. The active ingredient in CALAA-01 is a small interfering RNA (siRNA). This siRNA inhibits tumor growth via RNA interference to reduce expression of the M2 subunit of ribonucleotide reductase (R2). The CALAA-01 siRNA is protected from nuclease degradation within a stabilized nanoparticle targeted to tumor cells.

PURPOSE: This phase I trial will:

* Determine the safety, toxicity, and the maximum tolerated dose (MTD) of CALAA-01 when administered intravenously to patients with relapsed or refractory cancer.
* Characterize the pharmacokinetics (PK) of CALAA-01 after intravenous administration.
* Provide preliminary evidence of efficacy of intravenous CALAA-01 by evaluating tumor response.
* Recommend a dose of intravenous CALAA-01 for future clinical studies.
* Evaluate immune response, by measuring antibody and cytokine levels, and the effect of intravenous CALAA-01 on complement.

DETAILED DESCRIPTION:
CALAA-01 is a targeted nanocomplex that contains anti-R2 siRNA. The complete nanocomplex formulation consists of four components:

1. a duplex of synthetic, non-chemically-modified siRNA (C05C)
2. a cyclodextrin-containing polymer (CAL101),
3. a stabilizing agent (AD-PEG), and
4. a targeting agent (AD-PEG-Tf) that contains the human transferrin protein (Tf). The cationic polymer interacts electrostatically with anionic siRNA to assemble into nanocomplexes below approximately 100 nm in diameter that protect the siRNA from nuclease degradation in serum. The siRNA-containing nanocomplexes are targeted to cells that over express the transferrin receptor (TfR). Upon reaching a target cell, transferrin binds to TfRs on the cell surface and the siRNA-containing nanocomplex enters the cell by endocytosis. Inside the cell, chemistry built into the polymer achieves unpackaging of the siRNA from the nanocomplex, permitting it to function via RNA interference.

ELIGIBILITY:
Inclusion Criteria include:

* Subjects must be at least eighteen (18) years of age.
* Subjects must have the following:

  * Histologically- or cytologically-confirmed solid malignancy that is measurable or non-measurable recurrent or metastatic disease (i.e., evaluable; e.g., cytologically or radiologically-detectable disease, markers, etc.)
  * Measurable disease is metastatic or unresectable
  * Standard curative or palliative measures do not exist, are no longer effective, or are unlikely to be effective.
* Subjects must have tumors that have recurred after previous surgery and/or radiation.
* Subjects must have received prior adjuvant, neoadjuvant, or any other therapy for metastatic disease. No restriction is placed on the number of cycles or regimens of prior therapy.
* Subjects must have fully recovered from diagnostic or therapeutic surgery (i.e., complete wound healing).
* Subjects must have fully recovered from prior radiotherapy for local symptom palliation.
* Subjects must have recovered from the toxic effects of prior therapy.
* Women and men of child-bearing/conceiving potential must be willing to use highly effective contraceptive methods during the course of the study. Any female who is not sexually active must agree to begin using highly effective contraceptive methods if she becomes sexually active during the study. Females who are post-menopausal (i.e., no longer menstruating) must have been so for two (2) years.
* Females of child-bearing potential (e.g., not surgically sterilized or two (2) years post-menopausal) must have a negative urine pregnancy test at screening. Positive tests will be confirmed serologically.
* Subjects must have adequate marrow, hepatic, and renal function at the time of screening,.
* Subjects must be willing and able, in the opinion of the Investigator, to comply with the protocol tests and procedures.
* Subjects must be willing and able to give written informed consent.

Exclusion Criteria include:

* Pregnant or nursing females.
* Clinically-evident (e.g., abdominal distention, bulging and/or fluid wave) ascites or Grade 3 peripheral edema.
* Allergy(ies) to contrast media required for protocol testing.
* History of significant weight loss within four (4) weeks prior to baseline.
* Evidence of active, uncontrolled infection or unstable or severe intercurrent medical conditions.
* Peripheral venous access insufficient to permit infusion of intravenous CALAA-01 and acquisition of laboratory specimens.
* Alcoholism (dependency), alcohol or substance abuse within twelve (12) months prior to screening that has caused health consequences.
* Immunocompromised subjects, subjects with known autoimmune conditions, active hepatitis or human immunodeficiency virus (HIV) seropositivity.
* Prior gene transfer therapy or prior therapy with a cytolytic virus of any type.
* Any electrocardiogram (ECG) abnormality at screening documented by the Principal Investigator as clinically significant.
* Vaccinations of any kind within thirty (30) days of baseline.
* Use of any investigational agent or device within thirty (30) days of CALAA-01 administration.
* Any concomitant medical or psychiatric condition or social situation that would make it difficult to comply with protocol requirements.
* Subjects requiring anticonvulsants.
* Radiotherapy, cytotoxic chemotherapy, biologic, hormonal or immunotherapy or bone marrow transplantation within four (4) weeks of baseline; nitroureas within six (6) weeks. Current use of growth factors.
* A myocardial infarction within six (6) months prior to enrollment or having New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, cardiomyopathy, severe uncontrolled ventricular arrhythmias, left bundle branch block, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities (e.g., Long QT interval, Torsade de Pointes).
* Poorly controlled hypertension
* Prior corticosteroids as anticancer therapy within seven (7) days of baseline.
* Active CNS metastases or currently receiving dexamethasone for CNS disease.
* Major surgery within four (4) weeks of baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To determine the tolerability, safety profile and maximum tolerated dose (MTD) of intravenous CALAA-01. | 3 months

SECONDARY OUTCOMES:
To characterize the pharmacokinetics (PK) of CALAA-01 after intravenous administration. | 3 Months
To determine preliminary efficacy of intravenous CALAA-01 by evaluating tumor response. | 3 months
To recommend an intravenous dose of CALAA-01 for future clinical studies. | 3 month
To evaluate immune response, by measuring antibody and cytokine levels, and effect of intravenous CALAA-01 on complement. | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Ribas, M.D., Principal Investigator — UCLA Jonsson Comprehensive Cancer Center; Anthony W Tolcher, M.D., Principal Investigator — START (South Texas Accelerated Research Therapeutics); Yun Yen, M.D., Ph.D., Principal Investigator — City of Hope National Medical Center
Locations (3):
- United States (3):
  - City of Hope National Medical Center, Duarte, California
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - START (South Texas Accelerated Research Therapeutics), San Antonio, Texas

REFERENCES:
- [Background] Heidel JD, Yu Z, Liu JY, Rele SM, Liang Y, Zeidan RK, Kornbrust DJ, Davis ME. Administration in non-human primates of escalating intravenous doses of targeted nanoparticles containing ribonucleotide reductase subunit M2 siRNA. Proc Natl Acad Sci U S A. 2007 Apr 3;104(14):5715-21. doi: 10.1073/pnas.0701458104. Epub 2007 Mar 22. PMID 17379663
- [Background] Heidel JD, Liu JY, Yen Y, Zhou B, Heale BS, Rossi JJ, Bartlett DW, Davis ME. Potent siRNA inhibitors of ribonucleotide reductase subunit RRM2 reduce cell proliferation in vitro and in vivo. Clin Cancer Res. 2007 Apr 1;13(7):2207-15. doi: 10.1158/1078-0432.CCR-06-2218. PMID 17404105
- [Background] Bartlett DW, Davis ME. Impact of tumor-specific targeting and dosing schedule on tumor growth inhibition after intravenous administration of siRNA-containing nanoparticles. Biotechnol Bioeng. 2008 Mar 1;99(4):975-85. doi: 10.1002/bit.21668. PMID 17929316
- [Background] Heidel JD. Linear cyclodextrin-containing polymers and their use as delivery agents. Expert Opin Drug Deliv. 2006 Sep;3(5):641-6. doi: 10.1517/17425247.3.5.641. PMID 16948559
- [Result] Davis ME, Zuckerman JE, Choi CH, Seligson D, Tolcher A, Alabi CA, Yen Y, Heidel JD, Ribas A. Evidence of RNAi in humans from systemically administered siRNA via targeted nanoparticles. Nature. 2010 Apr 15;464(7291):1067-70. doi: 10.1038/nature08956. Epub 2010 Mar 21. PMID 20305636
- See also: Calando Pharmaceuticals Website — http://www.calandopharma.com/